CLINICAL TRIAL: NCT05623878
Title: 68Ga-labeled NY108 PET Imaging in Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Principal Investigator, Chunjing Yu, Director, Affiliated Hospital of Jiangnan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LS2020005
Record Dates: First submitted 2022-11-15; First posted 2022-11-21 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Prostatic Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-Anti-PSMA mAbs (Experimental)
  Interventions: Drug: 68Ga-labeled NY108

INTERVENTIONS:
Drug: 68Ga-labeled NY108 — Patients will receive a tracer (20-40mcg, IV) dose of 68Ga (2-5mCi) labelled NY108.

SUMMARY:
This is a single arm study to evaluate the safety and biodistribution of 68Ga-labeled NY108 (68Ga-NY108) PET Imaging in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily signed informed consent;
2. Age 18-75, male;
3. Patients diagnosed with prostatic cancer confirmed by histopathology or cytology;
4. At least one measurable solid lesion has been examined according RECIST1.1 standard;
5. Patients with biopsy-proven PSMA positive;
6. ECOG score 0~3; Life expectancy of at least 3 months;

Exclusion Criteria:

1. Recovery from major trauma (including surgery) within 4 weeks prior to study treatment;
2. Patients with systemic or locally severe infections, or other serious coexisting diseases;
3. Patients with allergies or allergies to any component of the imaging agent or antibody;
4. Patients who cannot perform PET/CT imaging scan;
5. Patients with abnormal immune function or who have recently used immunosuppressive or potentiating agents including various vaccines;
6. Patients with autoimmune diseases, including rheumatoid arthritis; Inadequate control of arrhythmias, including atrial fibrillation;
7. Uncontrolled hypertension;
8. Syphilis, HBV, HCV, or HIV positive subjects;
9. Male subjects of reproductive age cannot take effective contraceptive measures;
10. Patients with a history of mental illness or related conditions;
11. Other subjects considered unsuitable by researchers.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of tissue distribution of 68Ga-Anti-PSMA mAbs(NY108) | 1 year
  Biodistribution of 68Ga-Anti-PSMA mAbs(NY108) evaluated by radioactive uptake values (standardized uptake values, SUVs) in various organs during repeated 68Ga-PET scans will be reported.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 1 year
  Safety will be assessed by evaluation of incidence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Chunjing Yu, Principal Investigator — Affiliated Hospital of Jiangnan University
Locations (1):
- Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fu H, Lou K, He H, Wang Y, Mi Y, Li W, Chen L, Zhang Y, Yu C. A novel PSMA targeted dual-function near-infrared fluorescence and PET probe for the image-guided surgery and detection of prostate cancer. Eur J Nucl Med Mol Imaging. 2024 Aug;51(10):2998-3008. doi: 10.1007/s00259-023-06492-x. Epub 2023 Nov 2. PMID 37914976